CLINICAL TRIAL: NCT04072666
Title: Investigations of Psychological Interventions in Suicide Prevention: A Comparison of Brief Cognitive Behavioural Therapy and the Attempted Suicide Short Intervention Program
Brief Title: A Comparison of Brief Cognitive Behavioural Therapy (CBT) and the Attempted Suicide Short Intervention Program
Acronym: ASSIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gold Coast Hospital and Health Service (Other Government)
Collaborators: Bond University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APP1164644
Record Dates: First submitted 2019-08-08; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Suicide, Attempted
Keywords: Suicide Prevention; Suicide Attempt; Brief Intervention
MeSH Terms: conditions — Suicide, Attempted; Suicide Prevention | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomisation will occur after recruitment. Participants will be randomised to either SPP, SPP alone + ASSIP or SPP + CBT. An intent-to-treat approach will be used and all participants randomly assigned to treatment groups using the ralloc command of Stata, which will employ block randomisation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the clear differences in interventions, participants and those administering the interventions will not be blinded. However, those analysing data and assessing the outcomes will be blinded to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASSIP plus SPP (Experimental): Participants in the ASSIP group will receive a combination of the comprehensive clinical SPP (i.e. standardised assessment, risk evaluation and formulation, safety planning and follow-up), and the ASSIP psychological intervention where they will receive three therapy sessions followed by regular ongoing contact through individually focused letters sent over 24 months.
  Interventions: Behavioral: Attempted Suicide Short Intervention Program (ASSIP); Behavioral: Suicide Prevention Pathway (SPP)
- CBT plus SPP (Experimental): Participants in the CBT group will receive a combination of the comprehensive clinical SPP (i.e. standardised assessment, risk evaluation and formulation, safety planning and follow-up), and the CBT psychological intervention where they will receive five CBT 60-minute individual sessions.
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT); Behavioral: Suicide Prevention Pathway (SPP)
- SPP alone (Active Comparator): The Suicide Prevention Pathway (SPP) comprises seven steps:
  i) Initial screening - persons experiencing suicide ideation and who may also have a history of, or recent, suicide attempt, are placed on the pathway; ii) Assessment of suicide risk iii) Formulation of suicide risk (based on a prevention oriented approach) iv) Safety planning (collaboratively developed with the client) and Counselling on access to lethal means v) Structured follow-up (within 24-48 hrs); vi) Transition of care plan; and vii) Caring contacts - ongoing contact/support for the person for the next 2 years (through personalised letters or phone texts).
  Interventions: Behavioral: Suicide Prevention Pathway (SPP)

INTERVENTIONS:
Behavioral: Attempted Suicide Short Intervention Program (ASSIP) — The first session is based on a narrative interview with the consumer relating the personal story of how the point of attempting suicide was reached, videorecorded with consent. The second session involves the therapist and consumer watching the session together to reactivate the consumer's mental state during the crisis in a safe environment. Automatic thoughts, emotions, psychological pain and stress, and contingent behaviour are discussed. A psycho-educative handout is given to consumers. The third session involves discussing the handout. A credit card size leaflet is provided, with long term goals, individual warning signs and safety strategies listed, in addition to a card with crisis phone numbers. The sessions are followed by letters sent over 24 months (Michel, Valach & Gysin-Maillart, 2017).
  Arms: ASSIP plus SPP
Behavioral: Cognitive Behavioural Therapy (CBT) — The intervention incorporates skills development and emphasises internal self-management. Therapy focuses on the identification of internal, external and/or thematic triggers for suicidal thinking and behaviours, as well as factors that maintain the desire to suicide, using thought records and/or chain analyses. Therapy aims to challenge distortions and misconceptions, including core beliefs that interfere with the motivation to initiate the process of problem solving and distress tolerance, by working on acceptance of emotional and/or physical pain. The final phase of treatment focuses on relapse prevention. CBT can challenge maladaptive beliefs, improve problem solving skills and social competence.
  Arms: CBT plus SPP
Behavioral: Suicide Prevention Pathway (SPP) — The standardised care approach involves a Suicide Prevention Pathway (SPP) modelled on the Zero Suicide Framework, utilising comprehensive chronological assessment of suicide events (CASE) (Shea, 2009) to elicit suicidal intent, the prevention orientated risk formulation (Pisani, Murrie, & Silverman, 2016), brief interventions conducted with the consumer during their initial assessment prior to the treatment setting (Stanley et al., 2016), Safety Planning Intervention, Counselling on Access to Lethal Means (CALM), brief patient/carer information, rapid, structured follow up, safe transitions of care and caring contacts (Fleischmann et al., 2008). The SPP is supported by a blended learning course with online and face-to-face training for staff.

SUMMARY:
The aim of this project is to assess if adding one of two structured suicide specific psychological interventions to a standardised clinical care approach improves outcomes for consumers presenting to a Mental Health Service with a suicide attempt.

The standardised care approach involves a Suicide Prevention Pathway (SPP) modelled on the Zero Suicide Framework.

The Attempted Suicide Short Intervention Program (ASSIP) is a manualised therapy composed of three therapy sessions following a suicide attempt, with subsequent follow up over two years with personalised mailed letters. Cognitive Behavioural Therapy (CBT)-Based Psychoeducational Intervention is a manualised approach involving brief CBT for suicide in five 60 minute sessions. The intervention incorporates skills development and emphasises internal self-management.

We will compare outcomes for:

1. The Attempted Suicide Short Intervention Program (ASSIP) + SPP, versus SPP alone
2. Five Sessions of Cognitive Behavioural Therapy (CBT) + SPP, versus SPP alone
3. CBT + SPP versus ASSIP + SPP.

Hypotheses:

1. The use of suicide specific psychological interventions (ASSIP; CBT) combined with a comprehensive clinical suicide prevention pathway (SPP) will have better outcomes than the clinical suicide prevention pathway alone.
2. Outcomes for the ASSIP + SPP and CBT + SPP will significantly differ.
3. Cost-benefit analyses will significantly differ between ASSIP and CBT.

DETAILED DESCRIPTION:
Key literature: Treatment approaches for suicide: The efficacy of various suicide prevention interventions has been the subject of research for some time, and includes a number of recent systematic reviews (e.g. Zalsman et al., 2016), and Gould, Greenberg, Velting, and Shaffer (2003) reviewed suicide prevention strategies specifically used with young people. Current national suicide prevention programs have highlighted the knowledge that suicide is a behaviour that stems from a complex and multifaceted set of circumstances and individual characteristics. These factors can be present across the human lifespan and occur across multiple cultural and community settings. The complex heterogeneous nature of the factors influencing suicide rates requires a collaborative and coordinated systems approach, incorporating strategies simultaneously implemented across multiple levels, including service systems, individualised interventions and community prevention. Despite this recognition, there remains a significant gap in the evidence base regarding the most effective interventions for use with suicide at the hospital service level.

In 2015, the Gold Coast Mental Heath and Specialist Services (GCMHSS) undertook a review of frameworks for suicide prevention to guide planning and choice of interventions, as well as enhancing the capability of the service and staff to provide interventions aimed at addressing the needs of people presenting as a result of a suicide attempt. Interventions were sought with available evidence of efficacy, based on outcomes obtained in clinical, controlled trials (particularly those suitable for the top six diagnostic related groups for mental health presenting to the Gold Coast Hospital Health Service (GCHHS), with the aim to provide recommendations for service wide implementation. The top six high priority mental health diagnostic groups included: schizophrenia & related disorders, mood/affective disorders, alcohol & substance related disorders, personality disorders, suicidal behaviours, and stress/adjustment/situational crisis. Two of the interventions that demonstrated the strongest quality of evidence included the Attempted Suicide Short Intervention Program (ASSIP) and Cognitive Behavioural Therapy (CBT) based psychological intervention.

This is a randomised controlled trial, with blinding of those assessing the outcomes.

Primary outcome measures: Representation to hospital with suicide attempt and/or suicidal ideations within 7, 14, 30 and 90 days post intervention. Death by suicide rates will also be examined. Death clearly assessed as not involving self-harm will be represented as not completing the study.

Secondary outcome measures: Self-reported level of suicidality, depression, anxiety, stress, resilience, problem solving skills and self- and therapist-reported level of therapeutic engagement.

Cost-benefit measures are assessed for both interventions.

All consumers who attempt suicide during the trial period, and are 16 years of age and older, will be offered the opportunity to join the trial. Specific demographic questions will identify the numbers of people who fall within specific target groups to enable a determination regarding any differences in the results being statistically significant.

A consumer/carer representative will participate on the research team, to inform the research and ensure sensitivity to the experiences of consumers with lived experience.

ELIGIBILITY:
Inclusion Criteria:

* Consumers aged 16 years and above residing in the Gold Coast catchment area
* Presenting to the Gold Coast Hospital with a recent suicide attempt and then placed on the Suicide Prevention Pathway.

Exclusion Criteria:

* Refusal of, or inability to, consent
* People who are already receiving specialised psychological interventions (such as CBT) will be excluded due to the potential confounding effect, but not people taking psychotropic medication

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 411 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Re-presentation to hospital with suicide attempt and/or suicidal ideations | 7 days post intervention
  Re-presentations to hospital emergency department (ED) with suicide attempts and/or suicidal ideations will be examined post intervention
Re-presentation to hospital with suicide attempt and/or suicidal ideations | 14 days post intervention
  Re-presentations to hospital emergency department (ED) with suicide attempts and/or suicidal ideations will be examined post intervention
Re-presentation to hospital with suicide attempt and/or suicidal ideations | 30 days post intervention
  Re-presentations to hospital emergency department (ED) with suicide attempts and/or suicidal ideations will be examined post intervention
Re-presentation to hospital with suicide attempt and/or suicidal ideations | 90 days post intervention
  Re-presentations to hospital emergency department (ED) with suicide attempts and/or suicidal ideations will be examined post intervention
Death by suicide rates | 24 months post intervention
  Death by suicide rates will also be examined post intervention

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline (pre-intervention); end of intervention (up to 5 weeks); and 6-, 12- and 24 months from baseline
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a suicide ideation and behaviour rating scale that supports suicide assessment through a series of simple, plain-language questions that anyone can ask. The maximum suicidal ideation category (1-5 on the C-SSRS) present at the assessment. A score of 0 indicates that no suicide ideation is present.
Depression, Anxiety and Stress Scale (DASS) | Baseline (pre-intervention); end of intervention (up to 5 weeks); and 6-, 12- and 24 months from baseline
  The Depression, Anxiety and Stress Scale (DASS) is a set of three self-report scales (21 item version) designed to measure the negative emotional states of depression, anxiety and stress. For this short (21-item) version of the DASS, Stress, Anxiety, and Depression scores a multiplied by 2 to get a score of 42 for each subscale (score 0-42). Higher scores of each subscale indicate higher emotional states of depression, anxiety, or stress.
The Coping Inventory for Stressful Situations (CISS) | Baseline (pre-intervention); end of intervention (up to 5 weeks); and 6-, 12- and 24 months from baseline
  The Coping Inventory for Stressful Situations (CISS) is a 48 item self-report questionnaire for clinical and non-clinical settings. The CISS is a four-factor model of human coping with adversity. The construct differentiates three types of coping: emotion-orientated (7 items), task orientated (7 items), and avoidance (distracted or social; 7 items). Respondents rate each item on a five point scale: (1) Not at all to (5) Very much. Scores range from 7-35 for each subscale (emotion-orientated coping, task-orientated coping, and avoidance coping). Higher scores indicate greater preference for task-orientated, emotion-orientated, or avoidance coping style.
Resilience Scale for Adults (RSA) | Baseline (pre-intervention); end of intervention (up to 5 weeks); and 6-, 12- and 24 months from baseline
  The Resilience Scale for Adults (RSA) is a 33 item self-report measure of resilience for adults. Items are rated on a 7-point scale: (1) Not true at all to (7) Very True. Higher scores indicate greater resilience (range 33 to 231).
Resilience Scale for Adolescents (READ) | Baseline (pre-intervention); end of intervention (up to 5 weeks); and 6-, 12- and 24 months from baseline
  The Resilience Scale for Adolescents (READ) is a 28 item self-report measure of resilience for adolescents. The scale consists of individual, family and external supports conceptual categories, and has been used to screen and profile for intervention. Items are rated on a 5-point scale: (1) Totally disagree (5) Totally agere. Higher scores indicate greater resilience (range 28 to 140).
The revised Helping Alliance Questionnaire - II (HAqII) | Baseline (pre-intervention); end of intervention (up to 5 weeks); and 6-, 12- and 24 months from baseline
  The revised Helping Alliance Questionnaire - II (HAqll) is a 19 item self-report questionnaire used to evaluate the quality of the patient-therapist relationship. Items are rated from (1) Strongly disagree to (6) Strongly agree. Total score ranges from 19 to 114. Higher scores indicate greater therapeutic alliance.
Independent-Interdependent Problem solving scale (IIPSS) | Baseline (pre-intervention); end of intervention (up to 5 weeks); and 6-, 12- and 24 months from baseline
  The Independent-Interdependent Problem solving scale (IIPSS) is a 10-item scale that measures dispositional preferences for independent and interdependent problem-solving. Items are rated from (1) Strongly disagree to (7) Strongly agree. Total score ranges from 10-70. Higher scores indicate greater preference for either independent or interdependent problem-solving style.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Stapelberg, MD, Principal Investigator — Gold Coast Health and Bond University; Kathryn Turner, MD, Principal Investigator — Gold Coast Health; Sabine Woerwag-Mehta, MD, Principal Investigator — Gold Coast Health and Bond University; Sarah Walker, Psy.D, Principal Investigator — Gold Coast Health; Anthony Pisani, Ph.D, Principal Investigator — University of Rochester; Konrad Michel, MD, Principal Investigator — Bern University Hospital
Locations (1):
- Gold Coast Hospital Health, Gold Coast, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pisani AR, Murrie DC, Silverman MM. Reformulating Suicide Risk Formulation: From Prediction to Prevention. Acad Psychiatry. 2016 Aug;40(4):623-9. doi: 10.1007/s40596-015-0434-6. Epub 2015 Dec 14. PMID 26667005
- [Background] Stanley B, Chaudhury SR, Chesin M, Pontoski K, Bush AM, Knox KL, Brown GK. An Emergency Department Intervention and Follow-Up to Reduce Suicide Risk in the VA: Acceptability and Effectiveness. Psychiatr Serv. 2016 Jun 1;67(6):680-3. doi: 10.1176/appi.ps.201500082. Epub 2016 Feb 1. PMID 26828397
- [Background] Bridge JA, Horowitz LM, Campo JV. ED-SAFE-Can Suicide Risk Screening and Brief Intervention Initiated in the Emergency Department Save Lives? JAMA Psychiatry. 2017 Jun 1;74(6):555-556. doi: 10.1001/jamapsychiatry.2017.0677. No abstract available. PMID 28456131
- [Background] Fleischmann A, Bertolote JM, Wasserman D, De Leo D, Bolhari J, Botega NJ, De Silva D, Phillips M, Vijayakumar L, Varnik A, Schlebusch L, Thanh HT. Effectiveness of brief intervention and contact for suicide attempters: a randomized controlled trial in five countries. Bull World Health Organ. 2008 Sep;86(9):703-9. doi: 10.2471/blt.07.046995. PMID 18797646
- [Background] Hassanian-Moghaddam H, Sarjami S, Kolahi AA, Lewin T, Carter G. Postcards in Persia: A Twelve to Twenty-four Month Follow-up of a Randomized Controlled Trial for Hospital-Treated Deliberate Self-Poisoning. Arch Suicide Res. 2017 Jan 2;21(1):138-154. doi: 10.1080/13811118.2015.1004473. Epub 2015 Mar 16. PMID 25774646
- [Background] Gysin-Maillart A, Schwab S, Soravia L, Megert M, Michel K. A Novel Brief Therapy for Patients Who Attempt Suicide: A 24-months Follow-Up Randomized Controlled Study of the Attempted Suicide Short Intervention Program (ASSIP). PLoS Med. 2016 Mar 1;13(3):e1001968. doi: 10.1371/journal.pmed.1001968. eCollection 2016 Mar. PMID 26930055
- [Background] Gysin-Maillart AC, Soravia LM, Gemperli A, Michel K. Suicide Ideation Is Related to Therapeutic Alliance in a Brief Therapy for Attempted Suicide. Arch Suicide Res. 2017 Jan 2;21(1):113-126. doi: 10.1080/13811118.2016.1162242. Epub 2016 Mar 16. PMID 26984644
- [Background] Michel K, Valach L, Gysin-Maillart A. A Novel Therapy for People Who Attempt Suicide and Why We Need New Models of Suicide. Int J Environ Res Public Health. 2017 Mar 1;14(3):243. doi: 10.3390/ijerph14030243. PMID 28257071
- [Background] Mayer KH, Bradford JB, Makadon HJ, Stall R, Goldhammer H, Landers S. Sexual and gender minority health: what we know and what needs to be done. Am J Public Health. 2008 Jun;98(6):989-95. doi: 10.2105/AJPH.2007.127811. Epub 2008 Apr 29. PMID 18445789
- [Background] Sanchez JP, Hailpern S, Lowe C, Calderon Y. Factors associated with emergency department utilization by urban lesbian, gay, and bisexual individuals. J Community Health. 2007 Apr;32(2):149-56. doi: 10.1007/s10900-006-9037-1. PMID 17571527
- [Background] De Leo D, Cerin E, Spathonis K, Burgis S. Lifetime risk of suicide ideation and attempts in an Australian community: prevalence, suicidal process, and help-seeking behaviour. J Affect Disord. 2005 Jun;86(2-3):215-24. doi: 10.1016/j.jad.2005.02.001. PMID 15935241
- [Background] Bennewith O, Evans J, Donovan J, Paramasivan S, Owen-Smith A, Hollingworth W, Davies R, O'Connor S, Hawton K, Kapur N, Gunnell D. A contact-based intervention for people recently discharged from inpatient psychiatric care: a pilot study. Arch Suicide Res. 2014;18(2):131-43. doi: 10.1080/13811118.2013.838196. PMID 24673299
- [Background] Bickley H, Hunt IM, Windfuhr K, Shaw J, Appleby L, Kapur N. Suicide within two weeks of discharge from psychiatric inpatient care: a case-control study. Psychiatr Serv. 2013 Jul 1;64(7):653-9. doi: 10.1176/appi.ps.201200026. PMID 23545716
- [Background] Zalsman G, Hawton K, Wasserman D, van Heeringen K, Arensman E, Sarchiapone M, Carli V, Hoschl C, Barzilay R, Balazs J, Purebl G, Kahn JP, Saiz PA, Lipsicas CB, Bobes J, Cozman D, Hegerl U, Zohar J. Suicide prevention strategies revisited: 10-year systematic review. Lancet Psychiatry. 2016 Jul;3(7):646-59. doi: 10.1016/S2215-0366(16)30030-X. Epub 2016 Jun 8. PMID 27289303
- [Background] Gould MS, Greenberg T, Velting DM, Shaffer D. Youth suicide risk and preventive interventions: a review of the past 10 years. J Am Acad Child Adolesc Psychiatry. 2003 Apr;42(4):386-405. doi: 10.1097/01.CHI.0000046821.95464.CF. PMID 12649626
- [Background] Bryan CJ, Wood DS, May A, Peterson AL, Wertenberger E, Rudd MD. Mechanisms of Action Contributing to Reductions in Suicide Attempts Following Brief Cognitive Behavioral Therapy for Military Personnel: A Test of the Interpersonal-Psychological Theory of Suicide. Arch Suicide Res. 2018 Apr-Jun;22(2):241-253. doi: 10.1080/13811118.2017.1319313. Epub 2017 Jun 1. PMID 28422576
- [Background] Stanley B, Brown G, Brent DA, Wells K, Poling K, Curry J, Kennard BD, Wagner A, Cwik MF, Klomek AB, Goldstein T, Vitiello B, Barnett S, Daniel S, Hughes J. Cognitive-behavioral therapy for suicide prevention (CBT-SP): treatment model, feasibility, and acceptability. J Am Acad Child Adolesc Psychiatry. 2009 Oct;48(10):1005-1013. doi: 10.1097/CHI.0b013e3181b5dbfe. PMID 19730273
- [Background] Shea SC. The chronological assessment of suicide events: a practical interviewing strategy for the elicitation of suicidal ideation. J Clin Psychiatry. 1998;59 Suppl 20:58-72. PMID 9881539
- [Derived] Stapelberg NJC, Bowman C, Woerwag-Mehta S, Walker S, Davies A, Hughes I, Michel K, Pisani AR, Van Engelen H, Delos M, Hageman T, Fullerton-Smith K, Krishnaiah R, McDowell S, Cameron A, Scales TL, Dillon C, Gigante T, Heddle C, Mudge N, Zappa A, Edwards M, Gutjahr S, Joshi H, Turner K. A lived experience co-designed study protocol for a randomised control trial: the Attempted Suicide Short Intervention Program (ASSIP) or Brief Cognitive Behavioural Therapy as additional interventions after a suicide attempt compared to a standard Suicide Prevention Pathway (SPP). Trials. 2021 Oct 21;22(1):723. doi: 10.1186/s13063-021-05658-y. PMID 34674732
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617